CLINICAL TRIAL: NCT04594174
Title: Prediction Model of the Blood Pressure Response to the Administration of Fluids in Abdominal Surgery Using the Pram Method.
Acronym: PREDICTPRAM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Oscar Diaz-Cambronero, Anesthetist, Hospital Universitario La Fe
Other Study IDs: PREDICTPRAM V.2019-318-1
Record Dates: First submitted 2020-10-05; First posted 2020-10-20 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Open Abdominal Surgery
MeSH Terms: interventions — Hypodermoclysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responders
  Interventions: Procedure: Fluid administration
- Non responders
  Interventions: Procedure: Fluid administration

INTERVENTIONS:
Procedure: Fluid administration — Patients will be treated in accordance with the criteria of the responsible physician and the hemodynamic data obtained with the Mostcareup monitor will be recorded and used for decision-making according to the hemodynamic management protocols of each center.
  If the patient has a PPV ≥ 14%, for 3 minutes and a MAP <65 mm Hg or a Systolic Blood Pressure <90 mm Hg, a bolus volume load of 3 ml / kg weight of a balanced crystalloid solution in a time of 10 minutes36,37. The start of the volume charge (T1) will be noted by an event mark on the MostCareup monitor. The end of the volume charge (T2) will be noted by an event mark on the MostCareup monitor. Five minutes after the completion of the volume charge a new event will be marked on the MostCare monitor (T3). Both brands will serve as a reference for the analysis of hemodynamic data. Patients will be considered responders to the administration of fluids if the cardiac index (CI) increase.

SUMMARY:
Fluid therapy is considered a first-line therapy in resuscitation protocols for hemodynamically unstable patients. The administration of fluids usually translates into an increase in Cardiac Output. However, not all patients increase mean blood pressure after fluid administration.

To determine if fluids the administration improves blood pressure, it is necessary to evaluate the dependence of preload, vasomotor tone, and left ventricular stroke volume.

The aim of this study is to confirm the usefulness of dynamic elastance, cardiovascular impedance, cardiac cycle efficiency, and other hemodynamic parameters calculated with the PRAM method as predictors of blood pressure response after fluid administration in open abdominal surgery. This will allow us to make and evaluate a predictive model for the blood pressure response after fluid administration in open abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Patients scheduled for open abdominal surgery lasting ≥ 120 minutes under general anesthesia with mechanical ventilation and the use of VT of 8 ml / kg ideal weight and who require serious arterial monitoring.

Exclusion Criteria:

* Patients <18 years.
* Patients> 80 years.
* Pregnant women.
* Urgent surgery.
* ASA >3
* Pathologies that may alter the quality of the arterial signal due to alterations of the dicrotic incisura.
* Poor quality of the arterial pressure wave due to artifacts of the transduction system (resonance and damping).
* Personal history of:
* Cardiac arrhythmia.
* Left ventricular ejection fraction <30%
* Right ventricular dysfunction (peak systolic tricuspid annulus velocity <0.16 m / sec)
* Intracardiac shunt
* Preoperative creatinine> 1.4 mg / dl.
* Dialysis
* Previous treatment with beta-blockers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for open abdominal surgery, older than 18 years. All sex participates and not gender based.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Dynamic elastacy ratio PPV/SVV | During surgery
  PPV/SVV